CLINICAL TRIAL: NCT02106364
Title: A Comparison of LY2605541 Versus Insulin Glargine as Basal Insulin Treatment in Combination With Oral Anti-Hyperglycemia Medications in Insulin-Naïve Patients With Type 2 Diabetes Mellitus: An Open-Label, Randomized, 52-week Study
Brief Title: A Study of Insulin Peglispro (LY2605541) in Participants With Type 2 Diabetes Mellitus
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Lilly's decision to cancel this trial is due to regulatory uncertainty in China.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13564; I2R-MC-BIDB (Other: Eli Lilly and Company)
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2016-03-28 (Estimated); Status verified 2016-03

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — basal insulin peglispro; LY2605541; Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LY2605541 (Experimental): LY2605541 administered by subcutaneous (SQ) injection once daily for 52 weeks. Initial dose is 10 units (10 U) and is titrated by investigator. Participants may continue oral antihyperglycemic medication (OAM) as prescribed by their personal physician.
  Interventions: Drug: Insulin Peglispro
- Insulin Glargine (Active Comparator): Insulin glargine administered by SQ injection once daily for 52 weeks. Initial dose is 10 U and is titrated by investigator. Participants may continue OAM as prescribed by their personal physician.
  Interventions: Drug: Insulin Glargine

INTERVENTIONS:
Drug: Insulin Peglispro — Administered SQ
  Other Names: LY2605541
  Arms: LY2605541
Drug: Insulin Glargine — Administered SQ
  Arms: Insulin Glargine

SUMMARY:
The main purpose of this study is to compare the efficacy and safety of a new basal insulin, insulin peglispro, to insulin glargine in participants with type 2 diabetes mellitus (T2DM). Both drugs will be given by an injection under the skin. Participants may continue to take oral antihyperglycemic medication (OAM) during the study, as prescribed by their personal physician. The study is expected to last about 12 months for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Have T2DM (per World Health Organization [WHO] Classification of Diabetes) not treated with insulin.
* Have had diabetes for at least 1 year.
* Have been receiving at least 2 oral antihyperglycemic medications (OAMs) for at least 3 months prior to the study.
* Have hemoglobin A1c (HbA1c) of 7.0% to 11.0%, inclusive, according to central lab at screening.
* Have body mass index (BMI) ≤40 kilogram/square meter (kg/m^2).
* This inclusion criterion applies to females of child-bearing potential (not surgically sterilized and between menarche and 1-year postmenopausal) only: are not breastfeeding, test negative for a serum pregnancy test, intend not to become pregnant during study or willing to have a reliable method of birth control.

Exclusion Criteria:

* Insulin therapy: have used insulin therapy (outside of pregnancy) anytime in the past 2 years, except for short-term treatment of acute conditions, and up to a maximum of 4 continuous weeks. Insulin use of any duration during pregnancy is not considered an exclusion criterion.
* Concomitant medications: rosiglitazone, pramlintide, glucagon-like peptide-1 (GLP-1) receptor agonist (for example, exenatide, exenatide once weekly, or liraglutide) used concurrently or within 3 months prior to screening.
* Local OAM restrictions: for participants on OAMs, restrictions for cardiac, renal, hepatic diseases and maximum dose, local product regulations must apply.
* Weight loss medications: are currently taking, or have taken within the 3 months preceding screening, prescription or over-the-counter medications to promote weight loss.
* Severe hypoglycemia history: have had any episodes of severe hypoglycemia within 6 months prior to screening.
* Diabetic ketoacidosis (DKA) or hyperglycemic hyperosmolar nonketotic coma (HHNKC): have had 1 or more episodes of DKA or hyperosmolar state/coma in the past 6 months.
* Cardiovascular: have cardiac disease with functional status that is New York Heart Association Class III or IV (per New York Heart Association [NYHA] Cardiac Disease Classification).
* Renal: have a history of renal transplantation, or are currently receiving renal dialysis or have serum creatinine ≥2 milligram/deciliter (mg/dL) (177 micromole/liter [mol/L]).
* Hepatic: have obvious clinical signs or symptoms of liver disease (excluding non-alcoholic fatty liver disease [NAFLD]), acute or chronic hepatitis, non-alcoholic steatohepatitis (NASH), or elevated liver enzyme measurements.
* Lipid-lowering medications:

  * Are using niacin preparations as a lipid-lowering medication or bile acid sequestrants within 90 days prior to screening; or,
  * Are using lipid-lowering medication at a dose that has not been stable for ≥90 days prior to screening.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Hemoglobin A1c (HbA1c) at 26 Week Endpoint | Baseline, 26 Weeks

SECONDARY OUTCOMES:
Proportion of Participants with HbA1c ≤6.5% and <7.0% | Week 26 and Week 52
Proportion of Participants with HbA1c <7.0% Without Nocturnal Hypoglycemia Event | Baseline through 26 Weeks and Baseline through 52 Weeks
Rate of Total and Nocturnal Hypoglycemia Events | Baseline to 26 Weeks
Fasting Serum Glucose (FSG) by Laboratory Measurements | 26 Weeks
9 Point Self Monitored Blood Glucose | 26 Weeks
Change from Baseline in Body Weight at Week 26 Endpoint | Baseline, 26 Weeks
Change from Baseline in HbA1c at 52 Week Endpoint | Baseline, Week 52
Insulin Dose by Unit | 26 Weeks
Time to Reach Steady-State | Baseline through 52 Weeks
Fasting Blood Glucose by Self Monitoring | Baseline through 52 Weeks
Intra-Participant Variability in Fasting Blood Glucose | Baseline through 52 Weeks
Change from Baseline in EuroQol-5 Dimension Questionnaire (EQ-5D) Score | Baseline, Week 26, Week 52
Change from Baseline in the Low Blood Sugar Survey (LBSS) | Baseline, Week 26, Week 52
Number of Participants Developing Anti-Insulin Peglispro Antibodies | Week 26 and Week 52
Change from Baseline in Lipid Profile | Baseline, Week 26

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (10):
- United States (10):
  - Rheumatology Associates PC, Birmingham, Alabama
  - Florida Medical Clinic PA, Zephyrhills, Florida
  - Diagnostic Rheumatology and Research, Indianapolis, Indiana
  - Heartland Research Associates, Wichita, Kansas
  - Washington University Medical Center, St Louis, Missouri
  - Albuquerque Rehabilitation & Rheumatology, PC, Albuquerque, New Mexico
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Carolina Arthritis Associates, Wilmington, North Carolina
  - STAT Research, Dayton, Ohio
  - Apex Clinical Research, Kennewick, Washington